CLINICAL TRIAL: NCT05615077
Title: Effectiveness of Comprehensive Intervention for the Prevention of Fall in Older Adults; a Randomized Controlled Trial
Brief Title: Multidisciplinary Combined Exercise and Education Intervention for Falls in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Principal Investigator, Keewon Kim, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2208-176-1354
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Falls Prevention
Keywords: Falls, exercise, education, elderly
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined exercise-education intervention group (Experimental): Combined exercise-education intervention by fall risk state for 12 months during intervention period.
  Interventions: Other: Combined exercise-education intervention
- Control group (No Intervention): No intervention for 12 months during intervention period.

INTERVENTIONS:
Other: Combined exercise-education intervention — Combined exercise and education intervention by fall risk state for 12 months during intervention period.
  Exercise intervention includes balance exercise and strength exercise according to protocol.
  Education intervention includes medication review, nutrition intervention, and home hazard modification.
  The key to medication review is paying special attention to medications known to increase the risk of falls. Reduction of these medications is recommended, and redundant psychotropic medications are withdrawn. Nutrition intervention includes investigating dietary habits and calculate insufficient protein intake to provide customized diet and high protein drink. If vitamin D necessary, supplements are prescribed. Home hazard modification includes providing instructions to reduce and modify the home hazards that increase the risk of falls.
  Arms: Combined exercise-education intervention group

SUMMARY:
This study aims to demonstrate the effect of combined exercise-education intervention in old adults with fall risk. This study will be conducted with prospectively randomized controlled trial comparing outcome of combined exercise-education intervention with conventional medical care. Falls efficacy scale-international, fall history, Balance function, handgrip strength, gait speed, knee extensor muscle power, physical performance, muscle mass using DEXA and BIA, quality of life, depression, cognitive function, activities of daily living, nutritional assessment will be evaluated on baseline, 1-month, 3-months, 6-months, and 12-months after intervention.

DETAILED DESCRIPTION:
A fall is defined as an event which results in a person coming to rest inadvertently on the ground or floor or other lower level. And also, falls are the second leading cause of unintentional injury deaths worldwide. In particular, adults older than 65 years of age suffer the greatest number of fatal falls. It has been reported exercise in fall risk patients not only improved physical performance but also reduced the fall risk. Also, it is recently demonstrated that combined exercise-education (e.g., exercise training, medication review, nutrition counseling, home hazards modification) intervention reduced fall risk in elderly patients. However, there is still not established standard protocol for the combined exercise-education intervention. Therefore, the aim of this trial is to compare the effects of combined exercise-education intervention in fall risk patients with multicenter, multidisciplinary, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 65 years and under 90 years
* if at least one <3 key question> is met or <stay independent score> ≥ 4 points
* patients who can walk more than 10m without an assistive device (ambulatory without an assistive device)
* patients who are willing to participate in exercise intervention for 12 months
* patients who can receive information about this study, submit written consent before participating in the study, and can comply with the requirements of the clinical trial

Exclusion Criteria:

* medically unstable conditions (e.g., cirrhosis with complications, end-stage renal failure requiring regular dialysis, hemorrhagic disease, uncontrolled hypertension, those who have been treated for a malignant tumor within 5 years)
* in case of ongoing neurological deficit except for stroke survivors (e.g., dementia, Alzheimer's disease, Parkinson's disease, etc.)
* decreased cardiopulmonary function such as heart failure, chronic obstructive pulmonary disease
* musculoskeletal problems that affect physical function and athletic ability (e.g., those who have undergone hip joint surgery, artificial joint surgery, spine surgery within the last 1 year)
* patients who have experienced alcohol abuse within the last 1 year (if 3 or more are meet in Cut off, Annoyed, Guilty, Eye opener [CAGE] evaluation)
* in case the purpose of this clinical trial cannot be understood or the matters necessary for the study cannot be carried out
* when it is judged by other researchers that the subject's condition makes it difficult to participate in this study

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Korean Version of Falls Efficacy Scale-International (KFES-I) | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Change from baseline falls efficacy to 1, 3, 6, 12 months after assessment, measured by Korean Version of Falls Efficacy Scale-International (KFES-I) [range from 16 to 64]. A higher value represents a high concern for falling.

SECONDARY OUTCOMES:
Falls history & injury | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Evaluation of number of falls and type of falls in previous 12 months
Physical performance | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Short Physical Performance Battery [range from 0 to 12 score]
Gait speed test | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  measured by 10 meter gait speed
Balance function | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Evaluation of physical balance function using Mini-Balance Evaluation System Test (Mini-BESTest) [range from 0 to 28]. Low value means poor ability of balance function.
Handgrip strength | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  measured in kilograms (kg) using hand-held dynamometer
Knee extensor muscle test | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  measured using a belt-stabilized hand-held dynamometer
Physical activity volume | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Evaluation of physical activity volume using Korean version of Physical Activity Scale for the Elderly (K-PASE) [range from 0 to 360 score]. Low value means poor physical activity
Cognitive function | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Evaluation of cognitive function using Korean-Montreal Cognitive Assessment (K-MoCA) [range from 0 to 30 score]. Low value means poor cognitive function
Health related quality of life | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Evaluation of quality of life using EuroQol-5 dimension (EQ-5D) [range from 5 to 25 score]. Higher value means worse quality of life
Depression status | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Evaluation of depression status using Patient Health Questionnaire-9 (PHQ-9) [range from 0 to 27 score]. Higher score indicates a higher severity of depressive symptoms
Nutritional Assessment | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  Evaluation of nutritional state using Mini-Nutritional Assessment short form (MNA-SF) [range from 0 to 14 score]. Low value means poor nutrition status
Appendicular skeletal muscle mass | Baseline (visit 1), 1 month after intervention (visit 2), 3 months after intervention (visit 3), 6 months after intervention (visit 4), 12 months after intervention (visit 5)
  measured using Bioelectrical Impedance Analysis (BIA)
Bone density | Baseline (visit 1), 12 months after intervention (visit 5)
  measured using Dual-energy X-ray absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Keewon Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palvanen M, Kannus P, Piirtola M, Niemi S, Parkkari J, Jarvinen M. Effectiveness of the Chaos Falls Clinic in preventing falls and injuries of home-dwelling older adults: a randomised controlled trial. Injury. 2014 Jan;45(1):265-71. doi: 10.1016/j.injury.2013.03.010. Epub 2013 Apr 8. PMID 23579066